CLINICAL TRIAL: NCT03560427
Title: Duloxetine Potentiates the Analgesic Efficacy of Intrathecal Morphine in Major Abdominal Cancer Surgery
Brief Title: Duloxetine Potentiates the Analgesic Efficacy of Intrathecal Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, lecturer of anesthesia and pain management , Assuit university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563-534
Record Dates: First submitted 2018-05-19; First posted 2018-06-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- duloxetine+morphine (Experimental)
  Interventions: Drug: Duloxetine 60mg
- placebo+morphine (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine 60mg — Patients will receive duloxetine, 60 mg tablet 2 hour before operation and will be anesthetized by combined spinal-general anesthesia that includes: spinal anesthesia with morphine 0.3 mg delivered in L4-5 inter spinous space.
  General anethseia: Induction of anesthesia was done by intravenous fentanyl, 2 µg / kg and propofol 1 - 2 mg / kg. Endotracheal intubation was achieved by cis-atracurium, 0.15 mg / kg. Maintenance of anesthesia was done by isoflurane and cis-atracurium, 0.03 mg / kg on demand. Additional intraoperative analgesia was consisted of administration of intravenous boluses of fentanyl, 50 µg according to the attending anesthesiologist's decision. At the end of surgery, muscle relaxation was reversed using neostigmine 0.05 mg / kg and atropine 0.01 mg / kg.
  Arms: duloxetine+morphine
Drug: placebo — Patients will receive placebo tablet 2 hour before operation and will be anesthetized by combined spinal-general anesthesia that includes: spinal anesthesia with morphine 0.3 mg delivered in L4-5 inter spinous space.
  General anethseia: Induction of anesthesia was done by intravenous fentanyl, 2 µg / kg and propofol 1 - 2 mg / kg. Endotracheal intubation was achieved by cis-atracurium, 0.15 mg / kg. Maintenance of anesthesia was done by isoflurane and cis-atracurium, 0.03 mg / kg on demand. Additional intraoperative analgesia was consisted of administration of intravenous boluses of fentanyl, 50 µg according to the attending anesthesiologist's decision. At the end of surgery, muscle relaxation was reversed using neostigmine 0.05 mg / kg and atropine 0.01 mg / kg.
  Arms: placebo+morphine

SUMMARY:
Duloxetine is a serotonin-norepinephrine reuptake inhibitor primarily used for treatment of major depression and anxiety. Duloxetine also has been used in the treatment of chronic pain conditions, such as osteoarthritis and musculoskeletal pain. There are few studies examining its effect for acute pain. The objective of this study is to evaluate the analgesic effect of duloxetine combined with intrathecal morphine for patients subjected to major abdominal cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* adult patients, subjected to major abdominal cancer surgery

Exclusion Criteria:

* patients on chronic opioid therapy
* patients allergic to study drugs (duloxetine+morphine)
* patients have uncontrolled hypertension and or ischemic heart disease

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
time to first analgesic request | 48 hours postoperatively
  the time elapsed from (0 hour = immediately postoperative) to time of first demand to analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Diab Hetta, MD, Principal Investigator — Lectuere of anesthesia and pain management
Locations (1):
- Diab, Asyut, Assuit, Egypt